CLINICAL TRIAL: NCT05544578
Title: Korean Translation and Validation of the Household Emergency Preparedness Instrument (K- HEPI) by a Phase 1 Feasibility Study in New York City
Brief Title: Korean Translation and Validation of the K-HEPI in NYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0542-Hunter
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-10

CONDITIONS: Disaster; Vulnerable Populations
Keywords: immigrants; civil defense; hazard; emergency; preparedness; planning; readiness; kit; disaster planning; emergency preparedness; community; community nursing; health surveys; intervention study
MeSH Terms: conditions — Emergencies; Piebaldism

STUDY DESIGN:
Intervention Model Description: This is a phase 1 feasibility study via a cluster randomized controlled trial.
Who Masked: Participant
Masking Description: The data collection site will be the unit of randomization. The participants will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurses Taking On Readiness Measures (N-TORM) Intervention Group (Experimental): This is a phase 1 feasibility study via a cluster randomized controlled trial.
  Interventions: Behavioral: Nurses Taking On Readiness Measures (N- TORM)
- Disaster and Emergency Preparation Pocket Guide Control Group (No Intervention): The control group will receive the Korean version of the 2-page Prepared New York: Disaster and Emergency Preparation pocket guide (NYC Emergency Management, n.d.) after data collection has been completed.

INTERVENTIONS:
Behavioral: Nurses Taking On Readiness Measures (N- TORM) — The intervention group will be educated about household emergency preparedness via a presentation and the Korean version of a New York City community-specific booklet called Ready New York: My Emergency Plan (NYC Emergency Management, 2022). The intervention will begin with instructing the participant to start the booklet during class 1 and completing it for homework. The class content will complement the booklet and the K-HEPI. The booklet includes preparedness recommendations, evacuation zone information, a disaster supply kit contents list, local utility company contact information, shelter locations, and special needs and priority utility restoration registry information. During class 2, study personnel will check for completion of the booklets, answer any questions that the participants may have about the evacuation and communication plans and disaster kits, and facilitate group discussion to foster social support from other community members.
  Arms: Nurses Taking On Readiness Measures (N-TORM) Intervention Group

SUMMARY:
Nurses Taking on Readiness Measures (N-TORM) is an innovative nurse-driven household emergency preparedness intervention modeled after an existing community intervention provided by emergency management personnel. The proposed pilot studies will test the Korean translation of the Household Emergency Preparedness Instrument (K-HEPI) and describe the implementation and effectiveness of N-TORM in a community setting. The aims of this instrument translation study and cluster randomized controlled trial are to (a) field and pilot test the K-HEPI in order to perform psychometric testing on the instrument and generate reliability and validity data, (b) increase the accessibility of N-TORM to vulnerable populations, (c) evaluate the effectiveness of N-TORM to increase household emergency preparedness knowledge and behavior, (d) implement N-TORM in a community located in an area at increased risk for disasters, measuring consistency of delivery, time, and cost of N-TORM, and (e) describe the factors most necessary to maintain and expand N-TORM.

DETAILED DESCRIPTION:
The proposed instrument translation study will pilot test a Korean version of the Household Emergency Preparedness Instrument to perform psychometric testing on the instrument, generating reliability and validity data for an examination of cross-cultural equivalence.

Following the instrument translation study, the investigators will use the K-HEPI in a cRCT to measure the level of household emergency preparedness of an at-risk population before and after receiving the N-TORM intervention to measure intervention effectiveness and health impacts of an extreme weather event. The investigators will compare the intervention group's K-HEPI scores to the control group's K-HEPI scores at baseline, one-month follow up, and after an extreme weather event.

Hypotheses (H):

H1: The level of household emergency preparedness, as measured by the K-HEPI, will increase after an educational intervention.

H2: The K-HEPI will account for a significant proportion of the variance in emergency preparedness among the sampled Korean households.

H3: Households who participate in the N-TORM educational intervention will show significantly greater increases in household emergency preparedness, as measured by the K-HEPI, than households that do not participate in the intervention.

H 4.1: Factors commonly found to be predictors of household emergency preparedness will be significantly associated with post-test levels of household emergency preparedness both for participants who do (experimental group) and do not (control group) complete the intervention.

H 4.2: Factors commonly found to be predictors of household emergency preparedness will significantly interact with whether or not participants complete the intervention, such that barriers will affect those who do not complete the intervention more than they affect those who do complete it.

H 5.1: The inter-item reliability of the K-HEPI will be similar to that of the English version.

H 5.2: Confirmatory factor analysis will find a significant fit of the K-HEPI to the same factor structure of the items that is found in the English version.

H 5.2.1: Model fit indices for the Korean version will be similar to those of the English version.

Background:

Worldwide, extreme weather events and disasters continue to have devastating impacts on households, communities, and nations with increased morbidity, mortality, and infrastructural and economic devastation. Disasters are unforeseen events that overwhelm local capacity, often resulting in a request at the national or international level for external assistance. The Federal Emergency Management Agency, Centers for Disease Control, American Red Cross, and local government agencies have socially marketed the importance of household emergency preparedness for years, yet the US public largely remains unprepared for disasters. Although household emergency preparedness has not been empirically demonstrated to result in decreased disaster-related morbidity and mortality, it is plausible that self-sufficiency of households will result in disaster resilience. Families must prepare for conditions that all disasters create, regardless of geographical area or type of disaster, such as loss of electricity, water, and being unable to obtain supplies for several days due to the need for sheltering in place or disruptions in the supply chain. A household is considered prepared if members have created a family communication and evacuation plan and assembled a disaster kit containing enough food and water to sustain each member for at least one week.

In September 2021, due to Hurricane Ida flooding, at least 13 people died in New York City. Eleven died in their basement-level homes in Queens, and nearly all the victims were residents of Asian descent who lived in low-income Asian immigrant communities. According to the 2020 Census data, Asians represented about 14.3% of the population in New York City and 26% of Queens. Asians in New York City are more likely to be foreign born immigrants than other major racial groups. Undocumented immigrants are particularly vulnerable to social marginalization, low socioeconomic status, lack of societal resources, and limited English proficiency, resulting in difficulties seeking help during extreme weather events. However, Asian Americans' emergency preparedness has rarely been measured in disaster research. As a result of the experience of living through Hurricane Ida, members of the Asian immigrant community requested household emergency preparedness education and community interventions from members of the study team.

The study data can build evidence for a promising individual and community household emergency preparedness intervention. The effectiveness of N-TORM to increase household emergency preparedness knowledge and behavior can be evaluated so that the intervention may be revised and replicated within different populations. This intervention can also be used in longitudinal studies to determine whether there is an association between being prepared for a disaster and surviving the disaster without the need for rescue or outside assistance. For medically frail community members, it can be determined whether there is an association between being prepared for a disaster and surviving the disaster without an acute exacerbation of a chronic illness and with no change in baseline functional status.

Study Design: K-HEPI Translation and Field Testing

The HEPI will be translated and field tested according to the recommended instrument translation procedures of Feher Waltz et al., (2010, pp. 452-458) and Sperber (2004). The English to Korean translation will follow a symmetrical translation, utilizing a decentered process. This means both the source and target languages are considered equally important, with both versions of the instrument remaining loyal to meanings and open to revision. Investigators from two different cultures (US and South Korea) will collaborate on the translation.

Study Design: K-HEPI Pilot Testing and N-TORM Intervention

Once the final version of the translated HEPI is achieved, the instrument will be used in a cRCT study with the target population. The intervention versus control data collection sites will be the unit of randomization.

Only approved research personnel will be involved in the research procedures. The investigators are employed at Hunter College, the City University of New York, and their duties in this study will be conducted under their role as employees of Hunter College. In addition, Korean-speaking research assistants and community health workers will be hired and trained to assist with study procedures.

The intervention group will receive two, 1-hour, in-person classes to help them develop their family evacuation and communication plans, identify community resources, and assemble a disaster supply kit. Trained study personnel will use a lecture and the Korean version of a New York City community-specific booklet called Ready New York: My Emergency Plan as a handout to educate the participants about the essentials of household emergency preparedness. The control group will receive the Korean version of the 2-page Prepared New York: Disaster and Emergency Preparation pocket guide after data collection.

Recruitment Procedures. Potential K-HEPI Pilot Testing / N-TORM participants will be recruited from Korean Community Services of Metropolitan New York, Inc. (KCS).

Risks and Benefits. There is no more than minimal risk for participation in this study. Little to no feelings of discomfort are expected. There are no direct benefits to participating in this study. This research does not claim to present a therapeutic benefit to the participants. Participants who successfully complete the N-TORM intervention may be self-sufficient for up to 72-hours post-disaster, but the association between disaster preparedness level and disaster resilience has not been empirically tested. It is anticipated that this study will benefit society.

Intervention Fidelity. The principal investigator (PI) will educate the study team members on how to deliver the N-TORM intervention. Each study team member who will serve as an N-TORM instructor will demonstrate competency in intervention delivery by teaching back the intervention to the PI. The PI and study team will evaluate the N-TORM intervention delivery of each team member by providing praise and any necessary critique/corrective feedback after the practice session. All instructors will use the same presentation and booklet and will adhere to the study protocol methods. The PI or Site PI will observe at least one N-TORM session by each instructor to monitor intervention fidelity. The investigators will keep a record of how often the instructors met, what was covered, and length of time it took to deliver the intervention.

The N-TORM intervention will take place at faith- and community-based organizations affiliated with the Korean Community Services of Metropolitan New York, Inc. who agree to recruit participants and host the N-TORM intervention at their site. The participants' portion of the intervention will take place in their homes, between classes 1 and 2.

Data Analysis. Descriptive statistics of the sample will be reviewed prior to regression analyses examining the associations between the study variables. Hierarchical linear regression analyses with time nested in participants will be conducted. The change in the level of household emergency preparedness will be evaluated with the pre- and post-intervention scores on the K-HEPI. The improvement from pretest to posttest will be analyzed through repeated measures ANOVAs; the main goal of these ANOVAs is to test the effect of participation in the N-TORM intervention. However, one of the models will also include demographics covariates and variables measuring common facilitators and barriers to household emergency preparedness to test their effects on K-HEPI scores and the effectiveness of the intervention considering them. In addition, the change in score will be evaluated with a repeated measures matched pairs t-test. Finally, the mean household emergency preparedness pretest score for all the participants will be compared to the mean posttest score with a percentage change calculation.

The reliability of the HEPI will be measured by looking at the internal consistency of the items (ordinal α coefficients and item-total correlations). Confirmatory factor analysis using polychoric correlations will be used to examine the factor structure of the K-HEPI and to compare it with that of the English version. Known-group validity of the K-HEPI will be assessed by comparing the scores of the participants who self-reported that they were unprepared for a disaster before and after the N-TORM intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* 1 participant pr household
* understand and read Korean
* lives independently within the New York metropolitan area (i.e., not in a rehabilitation facility, long-term care facility, halfway house or prison)
* consents to participate

Exclusion Criteria:

* less than 18 years of age
* cognitive impairments
* Non-Korean speaking
* Non-Korean reading

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Korean Household Emergency Preparedness Instrument (K-HEPI) Score | through study completion, an average of 1 year
  The Korean Household Emergency Preparedness Instrument (K-HEPI) is an all-hazards, comprehensive, 51-question instrument used to ascertain if a respondent is prepared for disasters. Higher scores on the HEPI indicate higher levels of preparedness. Excluding the Access and Functional Needs (AFN) and Special Actions (SA) subscales that are not applicable to all respondents, the minimum score a participant could receive on the General Preparedness (GP) scale is 0 and the maximum score is 40 (1 point for each yes-response and 0 points for each no-response). There is support for face, content, and criterion validity of this instrument. The HEPI questions are objective and ask about what the respondent presently owns or does in a dichotomous format.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Heagele, PhD, RN, Principal Investigator — City University of New York, School of Public Health
Locations (1):
- Hunter College, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences (2nd ed.). Lawrence Erlbaum Associates.
- [Background] Cong, Z. & Chen, Z. (2022). How are Asian-Americans different from other races in disaster preparedness in the context of caregiving responsibilities and preparation information access?. Natural Hazards. https://doi.org/10.1007/s11069-022-05262-6
- [Background] Feher Waltz, C., Strickland, O. L., & Lenz, E. R. (2010). Measurement in nursing and health research (4th edition). Springer Publishing Company.
- [Background] Heagele TN, Adams LM, McNeill CC, Alfred DM. Validation and Revision of the Household Emergency Preparedness Instrument (HEPI) by a Pilot Study in the City University of New York. Disaster Med Public Health Prep. 2022 Mar 25;17:e126. doi: 10.1017/dmp.2022.35. PMID 35332858
- [Background] Heagele TN, McNeill CC, Adams LM, Alfred DM. Household Emergency Preparedness Instrument Development: A Delphi Study. Disaster Med Public Health Prep. 2022 Apr;16(2):570-582. doi: 10.1017/dmp.2020.292. Epub 2020 Nov 20. PMID 33213596
- [Background] Sperber AD. Translation and validation of study instruments for cross-cultural research. Gastroenterology. 2004 Jan;126(1 Suppl 1):S124-8. doi: 10.1053/j.gastro.2003.10.016. PMID 14978648
- [Background] Zheng G, Oksuzyan S, Hsu S, Cloud J, Jewell MP, Shah N, Smith LV, Frye D, Kuo T. Self-Reported Interest to Participate in a Health Survey if Different Amounts of Cash or Non-Monetary Incentive Types Were Offered. J Urban Health. 2018 Dec;95(6):837-849. doi: 10.1007/s11524-018-0237-7. PMID 29654397
- See also: Centre for Research on the Epidemiology of Disasters, United Nations Office of Disaster Risk Reduction (CRED-UNDRR) (2020). Human cost of disasters: 2000-2019. EM-DAT The international disaster database. — https://www.undrr.org/publication/human-cost-disasters-overview-last-20-years-2000-2019
- See also: Kriegstein, B., Parnell, W. Parisienne, T., Crane-Newman, M., Annese, J., Tracy, T., & McShane, L. (2021, September 2). Hurricane Ida NYC death toll rises to 13, including infant and senior citizen, after record rains and lethal flooding. New York Daily — https://www.nydailynews.com/new-york/nyc-crime/ny-hurricane-ida-rain-flooding-dead-20210902-moja6dep2renjlivacy3vyk6qi-story.html
- See also: NYC Emergency Management (n.d.). Guides and app. City of New York. — https://www1.nyc.gov/site/em/ready/guides-resources.page#myemergencyplan
- See also: United States Census Bureau (2021a, October 8). How ready are we? Measuring America's people, places, and economy. — https://www.census.gov/library/visualizations/2018/comm/how-ready-are-we.html
- See also: United States Census Bureau (2021b, November 15). 2020 census. — https://www.census.gov/programs-surveys/decennial-census/decade/2020/2020-census-main.html
- See also: Yam, K. & Venkatraman, S. (2021, October 18). Ida's forgotten victims: Nearly all storm's basement deaths were Asian residents, obscured by climate injustice. NBC News. — https://www.nbcnews.com/news/asian-america/ida-s-forgotten-victims-nearly-all-storm-s-basement-deaths-n1281670